CLINICAL TRIAL: NCT03013452
Title: A Randomized Controlled Trial of Long Term Airway Clearance With Oscillating Positive End Expiratory Pressure Device Versus Autogenic Drainage in People With Bronchiectasis
Brief Title: Oscillating PEP vs Autogenic Drainage in People With Bronchiectasis
Acronym: oPEP-vs-AD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carmel Medical Center (Other)
Collaborators: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMC-16-0087-CTIL
Record Dates: First submitted 2017-01-01; First posted 2017-01-06 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-02

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Intervention Model Description: 2 modes of physiotherapy: 1- autogenic drainage; 2- oscillating positive expiratory pressure device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Autogenic drainage (Active Comparator): Chest physiotherapy by autogenic drainage daily for 15 minutes each day, for 1 month. Instruction by a physiotherapist as to proper technique will be given at the beginning of the study.
  Interventions: Behavioral: Autogenic drainage
- oPEP (Active Comparator): Chest physiotherapy with an Aerobika oPEP device daily for 15 minutes each day for 1 month. Instruction by a physiotherapist as to proper technique will be given at the beginning of the study.
  Interventions: Device: oPEP

INTERVENTIONS:
Device: oPEP — Daily chest clearance (chest physiotherapy) using an oPEP (Aerobika) device.
  Other Names: Aerobika device
  Arms: oPEP
Behavioral: Autogenic drainage — Daily chest clearance (chest physiotherapy) by Autogenic Drainage method.
  Arms: Autogenic drainage

SUMMARY:
In this study, investigating two modes of chest physiotherapy on lung clearance index (LCI), 50 patients with bronchiectasis will be randomized to either oPEP or autogenic drainage.

DETAILED DESCRIPTION:
One of the fundamental treatments in the management of bronchiectasis is airway clearance, which effectively rids the airways of mucus to prevent secondary infection and inflammation. While effective airway clearance is widely accepted as a first line treatment, the choice of airway clearance method is complicated by lacking evidence base. One of the obstacles to establishing evidence of efficacy of an airway clearance technique or device is the limitations in the choice of endpoints.

Aerobika (Trudell medical international, Canada) is an oscillating positive expiratory pressure (oPEP) device, designed and developed for the effective clearance of secretions in people with suppurative lung diseases. It has been tested and found safe and effective in chronic obstructive pulmonary disease (COPD) - chronic bronchitis.

The lung clearance index (LCI) measured by multiple breath washout (MBW) is a measure of ventilation inhomogeneity and has been shown to be a sensitive lung function test in early lung disease. Its usefulness has been demonstrated in cystic fibrosis (CF), particularly in children and adults with mild disease. LCI has been assessed in bronchiectasis and has been found to be significantly different from normal subjects, and to correlate with Forced Expiratory Volume in 1 second (FEV1).

The aim of this study is to test the long term effect of daily lung clearance on LCI, quality of life and exacerbations using the Aerobika oPEP device versus autogenic drainage (AD) in people with bronchiectasis.

50 patients with confirmed bronchiectasis will be enrolled in this study. Participants will be randomized to daily physiotherapy with either Aerobika or Autogenic drainage. Change in LCI, measured before and after one month, will be the primary endpoint of this study.

ELIGIBILITY:
Inclusion Criteria:

1. High Resolution chest computerized tomography (HRCT) during stable disease imaging bronchiectasis in at least 2 lung lobes
2. Sputum production during most days of the year
3. Stable chronic therapy during last 4 weeks
4. FEV1 = 70% predicted or higher on spirometry
5. Able to give informed consent or assent
6. Age: 18- 80 years

Exclusion Criteria:

1. An exacerbation during last 4 weeks before randomization
2. Any change in respiratory medications during the past 4 weeks before randomization
3. A diagnosis of cystic fibrosis
4. A diagnosis of primary ciliary dyskinesia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-03-09 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in LCI | 1 month
  LCI will be determined before intervention and after 1 month and change will be recorded.

SECONDARY OUTCOMES:
Total score on QOL- B questionnaire | 1 month
  Patients will answer QOL-B questionnaire before and after 1 month of the intervention, and total score will be recorded.
Score on respiratory domain of QOL-B questionnaire | 1 month
  Patients will answer QOL-B questionnaire before and after 1 month of the intervention, and score on respiratory domain will be recorded.
FEV1 (% predicted)- difference from baseline | 1 month
  Spirometry will be performed before and after 1 month of the intervention, and change in FEV1 (% of predicted) will be recorded.
Forced Expiratory Volume (FVC) (% predicted)- difference from baseline | 1 month
  Spirometry will be performed before and after 1 month of the intervention, and change in FVC (% of predicted) will be recorded.

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Carmel Medical Center, Haifa
  - Pulmonology Institute, Carmel Medical Center, Haifa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flude LJ, Agent P, Bilton D. Chest physiotherapy techniques in bronchiectasis. Clin Chest Med. 2012 Jun;33(2):351-61. doi: 10.1016/j.ccm.2012.02.009. Epub 2012 Apr 4. PMID 22640850
- [Background] Robinson PD, Latzin P, Verbanck S, Hall GL, Horsley A, Gappa M, Thamrin C, Arets HG, Aurora P, Fuchs SI, King GG, Lum S, Macleod K, Paiva M, Pillow JJ, Ranganathan S, Ratjen F, Singer F, Sonnappa S, Stocks J, Subbarao P, Thompson BR, Gustafsson PM. Consensus statement for inert gas washout measurement using multiple- and single- breath tests. Eur Respir J. 2013 Mar;41(3):507-22. doi: 10.1183/09031936.00069712. Epub 2013 Feb 8. PMID 23397305
- [Result] Gonem S, Scadding A, Soares M, Singapuri A, Gustafsson P, Ohri C, Range S, Brightling CE, Pavord I, Horsley A, Siddiqui S. Lung clearance index in adults with non-cystic fibrosis bronchiectasis. Respir Res. 2014 May 18;15(1):59. doi: 10.1186/1465-9921-15-59. PMID 24884343
- [Result] Rowan SA, Bradley JM, Bradbury I, Lawson J, Lynch T, Gustafsson P, Horsley A, O'Neill K, Ennis M, Elborn JS. Lung clearance index is a repeatable and sensitive indicator of radiological changes in bronchiectasis. Am J Respir Crit Care Med. 2014 Mar 1;189(5):586-92. doi: 10.1164/rccm.201310-1747OC. PMID 24428575